CLINICAL TRIAL: NCT03282578
Title: Prospective Randomised Sternal Closure Study Sternalock 360 Plates vs Conventional Stainless Steel Wires
Brief Title: Sternalock Versus Wires for Sternal Closure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Colin Royse, Co-PI, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH 2017.165
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cardiac Surgery; Sternal Closure
Keywords: sternum; bone healing; recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sternalock 360 sternal plating system (Active Comparator): use of the SternaLock 360 system to close the sternum: 3 plates with 3 bands and measured screw length to engage but not penetrate the posterior sternal cortex, used to close the sternum
  Interventions: Device: Sternalock 360 sternal plating system
- Sternal wires (Active Comparator): Stainless steel sternal wires applied in a "figure of 8" configuration to close the sternum
  Interventions: Device: Sternal Wires

INTERVENTIONS:
Device: Sternalock 360 sternal plating system — The SternaLock 360 system is a band and plating system designed to improve sternal stability. 3 bands surround the sternum to oppose the bones (like wires), but an additional 3 plate system prevents anterior posterior displacement and provides a rigid fixation.
  Arms: Sternalock 360 sternal plating system
Device: Sternal Wires — Stainless steel wires are applied in a "figure of 8" configuration to close the sternum
  Arms: Sternal wires

SUMMARY:
Design:

Investigator Initiated Prospective Randomised Trial

Study Centre's:

Melbourne Private Hospital Royal Melbourne Hospital

Study Hypothesis:

Use of the SternaLock 360 will reduce the incidence of sternal motion > 2mm by absolute difference of 40% at 6 weeks of surgery compared to stainless steel wiring.

Use of the SternaLock 360 will improve bone healing and quality of recovery after surgery compared to stainless steel wiring

Study Objective:

To determine if the SternaLock 360 system reduces sternal instability, increases bone healing, and improves quality of recovery compared to stainless steel wiring of the sternum, after cardiac surgery involving median sternotomy

Inclusion Criteria:

Age ≥ 18 year old Elective cardiac surgery Primary cardiac surgical procedure No evidence of infection at time of surgery Sufficient English language to complete the Postoperative Quality of Recovery Survey

Exclusion Criteria:

Previous sternotomy (redo) Clinical sternal deformity Home locality preventing follow-up (e.g. remote regional, interstate or overseas patient)

Number of Planned Subjects:

50

DETAILED DESCRIPTION:
Introduction/Background Information Since the inception of cardiac surgery in the early 1960s, division of the sternum has provided the superior access to cardiac structures. Cardiac surgery may involve treatment of the coronary arteries, valves or major vessels such as the ascending aorta. In children, correction of congenital malformations is also performed.

The conventional bone fixation during the 1960s was the placement of stainless steel wires around or through the sternum, predominantly as single wires which were tensioned by twisting. In the 1980s, it became fashionable for some cardiac surgeons to pass the wire twice around the bone (as would be the case repairing a fence on a farm), so-called "figure of 8" configuration and tensioning again occurring by twisting the wires. There have been no adequate studies investigating which of these two techniques may be superior.

In simple terms, bone healing is promoted by

* Minimising movement of the bone edges at the fracture site and
* Improved alignment of the bone edges

The sternum is a connecting bone that moves in multiple planes to transfer load and position the limbs in space during every day functional tasks and respond to the demands of respiration. The healing of the sternum is in the context of many efforts by the treating physicians and physiotherapists to encourage activities that might cause distracting forces at the sternal fracture site. Additionally, simple everyday activities by the patient such as coughing, deep breathing, sneezing, transferring in and out of bed, turning over in bed and driving all lead to substantial distracting forces acting on the sternal fracture site1. External fixation is not encouraged because the patient needs to have significant chest wall movement in order to breathe and clear sputum as part of the recovery from surgery.

Also, ultrasound data suggests an additional mechanism by which sternal healing is compromised with conventional sternal wiring techniques. The shape of the sternum is complex 1. The upper part is called the manubrium to which the clavicles and first rib join, and is generally quite thick with a reasonably robust and cortex and strong marrow. By contrast, the body of the sternum which forms the majority of the sternum is thinner and the marrow is frequently less robust than for the manubrium. In both areas, the cortical bone is present superficially (anterior) and deep (posterior) with the marrow between. When sternal wires are used, and the two halves of the sternum brought together and tensioned by twisting the wires, best efforts made to ensure that the cortical bone edges on either side are opposed or well aligned (that is, that in the anterior and posterior direction that the two bone edges from either side of well opposed). Generally, this is quite well achieved, but not always. Yet, even with ultrasound studies performed 1 or 2 days after surgery, the alignment between the anterior cortical bone edge on either side is lost as detected by the cortical bone of one side overriding the cortical bone of the other side.

The implications of this ultrasound finding are twofold

1. Irrespective of the perfect alignment of the two sides of the sternal fracture at the time of surgery under general anaesthetic, coughing and deep breathing usually leads to distraction forces that results in one side of the divided sternum overriding the other side, typically by a couple of millimetres or so. This must be because there is less bone to bone force when the cortical bone edge is being forced against soft tissue or against the marrow than it would be if it were forced against the cortical bone of the other side. This is important because any distracting force caused by coughing or deep breathing or indeed any other activity should logically, result in the two halves of the sternal bone adopting a position of least force.
2. What this means is that the two halves of the sternum in combination (and after over riding has occurred) are now less wide than they had been at the time that the sternal wire was tensioned at the end of the surgical procedure, by the distance of the sternal override detected by the ultrasound.

Consequences of poor sternal healing: Patients may feel movement of the sternum and that may limit their activity. However, chronic sternal instability is associated with pain 2, which may in turn affect other aspects of daily living, require long term medications and predispose to depression.

SternaLock 360 system The SternaLock 360 system is a band and plating system designed to improve sternal stability. 3 bands surround the sternum to oppose the bones (like wires), but an additional 3 plate system prevents anterior posterior displacement and provides a rigid fixation. CT scan follow up shows improved bone healing at 3 months after surgery compared to conventional wires, but the CT scan is a poor measurement of dynamic movement. Quality of recovery and functional status has not been adequately studied.

The unique design of the SternaLock 360 system, is that it combines a

1. Compressive force to the two sternal halves forcing them together (similar to the principal of the sternal wires), thus counteracting lateral distracting forces.
2. Additionally, by the placement of metal plates that cross the fracture and are fixed on either side by screws, predominantly the plates acts to prevent anterior/posterior distracting forces; longitudinal translation and thus better maintain the cortical bone to cortical bone apposition between the two sides.

Pilot Data Our research group is experienced in assessing sternal motion with ultrasound 4. We have conducted sternal ultrasound measurements of sternal motion after surgery as part of clinical follow up.

Over all the SternaLock 360 results in a far greater rigid fixation as noted at the time of surgical implantation. Subsequent pilot ultrasound studies performed during dynamic distracting forces (such as coughing) reveal reduced or absent movement at the fracture site and better preservation of fracture alignment. Ultrasounds have been performed at varying intervals from Day 1 post-operative to 6 weeks post-operative, and ultrasounds of sternal wire fixation have been performed at varying intervals after 10 months post-operative. Our observations are that fewer than 10% of patients who have received the SternaLock 360 have had motion >2 mm, whereas patients with conventional wiring have motion > 2 mm in more than 50%.

Evidence Gap The SternaLock 360 is an effective system for closing the sternum. There are few comparative data investigating bone healing with CT scans, but the CT alone is a poor indicator of sternal instability. There is no long term comparative data on sternal micro motion, or quality of recovery outcomes to identify whether the SternaLock 360 system will improve patient centred outcomes over and above improved bone healing.

Study Objectives Hypothesis Use of the SternaLock 360 will reduce the incidence of sternal motion > 2mm by absolute difference of 40% at 6 weeks of surgery compared to stainless steel wiring.

Use of the SternaLock 360 will improve bone healing and quality of recovery after surgery compared to stainless steel wiring.

Study Aims To determine if the SternaLock 360 system reduces sternal instability, increases bone healing, and improves quality of recovery compared to stainless steel wiring of the sternum, after cardiac surgery involving median sternotomy.

Randomisation The randomization sequence will be produced using a computer generated randomization sequence, in unequal blocks. Concealment will be by placing the card containing the allocation information in double opaque sealed envelopes, and concealment will be maintained until after recruitment and the patients is admitted to the operating theatre. The treating surgical team will then open the envelopes to reveal the allocation after (1) weaning from cardiopulmonary bypass and (2) final confirmation from the treating surgeon that the patient is suitable to be randomised.

Statistical Methods Participants who are scheduled for cardiac surgery will be screened and recruited from the cardiac surgery operation lists, surgeon's clinics and pre-operative ward.

The initial contact will be made in person during the first contact session prior to surgery. In-patients scheduled for cardiac surgery will be screened on the ward.

Medical histories will be reviewed and screened for participant suitability and eligibility. Once the patient's medical history has been reviewed and the patient's eligibility has been confirmed, the patient is then approached by the research staff member and the process of informed consent will proceed.

Power Calculation and Study Size Sample size estimates are based on the primary outcome of sternal motion > 2 mm at any location at 6 weeks after surgery. From pilot data, fewer than 10% of patients who have received the SternaLock 360 have had motion >2 mm, whereas patients with conventional wiring have motion > 2 mm in more than 50%. Based on a Fischer's Exact test, Alpha of 0.05, power of 80% and two-tailed design, 25 participants are required in each group to detect a difference of 50% to 10% between groups, favoring the SternaLock 360 system. The sample size will increase to 26 in each group to account for an estimated 5% dropout rate. The total number will be 52 participants.

Statistical Methods To Be Undertaken The primary endpoint will be assessed using the Chi Squared test on the incidence of sternal motion > 2 mm at 6 weeks after surgery.

Postoperative Quality of Recovery Variables of "recovery" are dichotomized to "recovered" or "not recovered" based on whether they have returned to their baseline (preoperative) values or a better result than their preoperative values; at each of the time points when measurements are performed. A tolerance factor is included in the scoring of cognitive recovery to allow for performance variability 6. The secondary outcomes of recovery over time, analysis will be performed using the a general linear mixed model to investigate group differences over time.

Continuous data will be analyzed using independent samples t test, or repeated measures analysis of variance (RM ANOVA). A P[Symbol]0.05 will define statistical significance.

References

1. El-Ansary D, Waddington G, Adams R: Trunk stabilisation exercises reduce sternal separation in chronic sternal instability after cardiac surgery: a randomised cross-over trialAust J Physiother 2007; 53: 255-60
2. El-Ansary D, Waddington G, Adams R: Relationship between pain and upper limb movement in patients with chronic sternal instability following cardiac surgery. Physiother Theory Pract 2007; 23: 273-80
3. Nishimura T, Kurihara C, Sakano Y, Kyo S: Sternalock plating system for elderly post-sternotomy patients. J Artif Organs 2014; 17: 288-90
4. El-Ansary D, Waddington G, Adams R: Measurement of non-physiological movement in sternal instability by ultrasound. Ann Thorac Surg 2007; 83: 1513-6
5. Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ: Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology 2010; 113: 892-905
6. Royse CF, Newman S, Williams Z, Wilkinson DJ: A human volunteer study to identify variability in performance in the cognitive domain of the postoperative quality of recovery scale. Anesthesiology 2013; 119: 576-81

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year old Elective cardiac surgery Primary cardiac surgical procedure No evidence of infection at time of surgery Sufficient English language to complete the Postoperative Quality of Recovery Survey

Exclusion Criteria:

* Previous sternotomy (redo) Clinical sternal deformity Home locality preventing follow-up (e.g. remote regional, interstate or overseas patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Sternal motion | 6 weeks after surgery
  Sternal edge movement with coughing that is >2 mm in any location as measured by ultrasound (US)

SECONDARY OUTCOMES:
Sternal override | 1 day to 3 months
  Anterior/posterior displacement of the sternal edges
Sternal motion | 1 day to 3 months
  Sternal edge movement at rest and coughing that is >2 mm in any location as measured by ultrasound (US)
Lung ultrasound | 1 day to 3 months
  Lung ultrasound examination for pathology
Sternal wound infection | 1 day to 3 months
  Any deep or superficial wound infection
MACCE | 1 day to 3 months
  Major adverse cerebral and cardiac events
Sternal pain | 1 day to 3 months
  Visual analogue pain score
PostopQRS | 1 day to 3 months
  Postoperative Quality of recovery scale - a multidimensional scale to measure quality of recovery after surgery
FDQ | 1 day to 3 months
  Functional difficulty questionaire
Sternal closure time | 1 day to 3 months
  Time from commencement of passage of first wire or SternaLock band to time of completion of all wire tensioning or screw fixation in plates
Penetration of the posterior cortical bone by screws | 6-10 days after surgery
  Penetration of the posterior cortical bone by screws assessed by chest X-Ray
Degree of bone healing | 3 months
  Degree of bone healing by CT scan at 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Royse, MD, Principal Investigator — Melbourne Health
Locations (1):
- Melbourne Private Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Royse AG, El-Ansary D, Hoang W, Lui E, McCusker M, Tivendale L, Yang Y, Canty DJ, Royse CF. A randomized trial comparing the effects of sternal band and plate fixation of the sternum with that of figure-of-8 wires on sternal edge motion and quality of recovery after cardiac surgery. Interact Cardiovasc Thorac Surg. 2020 Jun 1;30(6):863-870. doi: 10.1093/icvts/ivaa040. PMID 32236553